CLINICAL TRIAL: NCT06841718
Title: Investigating the Neural Signature of Freezing of Gait Using Ambulatory Electroencephalography in Parkinson's Disease
Brief Title: Investigating the Neural Signature of Freezing of Gait in Parkinson's Disease
Acronym: FOG-EEG
Status: Enrolling by invitation | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Moran Gilat, Professor, KU Leuven
Other Study IDs: s69013
Record Dates: First submitted 2025-01-27; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Freezing of Gait; Basal Ganglia Diseases; Brain Disease; Movement Disorders; Neurodegenerative Disease
Keywords: Parkinson's Disease; electroencephalography (EEG); freezing of gait; gait problems
MeSH Terms: conditions — Parkinson Disease; Basal Ganglia Diseases; Brain Diseases; Movement Disorders; Neurodegenerative Diseases; Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Home assessment: All 28 participants will undergo a single home based assessment including a gait protocol as well as administering clinimetrics and questionnaires. Patients will be tested early in the morning after at least 12 hours without the anti-parkinsonian medication (= 'partial' OFF medication) and then about 1 hour after the intake of the first morning medication dose, when the subject reports reaching self-reported ON state (= ON medication). The gait protocol consist out of A) a trajectory in the participants home from the living room towards the bathroom and back, including a 360° turn as well as a figure-8 turn and going through a doorway and B) a daily living task. All tests will be conducted in a fixed order. The protocol will be conducted as a single task, with a dual task (serial subtraction task), with voluntary stops during different parts of the trajectory, and with an auditory cue (rhythm set 10% slower then typical cadence).

SUMMARY:
Freezing of Gait (FOG) is a disabling symptom of Parkinson's disease (PD) and a leading cause for falls. Current medical management is inadequate to alleviate FOG so there is need for improved treatments. A major draw-back in the development of better treatments for FOG is the difficulty in detecting episodes and our poor understanding of its underlying pathophysiology.

This study will investigate the cortical signature of FOG using ambulatory electroencephalography (EEG) to help improve FOG detection algorithms and provide novel insights into the underlying pathophysiology, which together will guide therapy development.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Parkinson's disease (PD) made by a Neurologist*
2. Modified Hoehn & Yahr (H&Y) Stage I to IV in the ON medication state
3. Age above 18 years*
4. Able to walk 5 minutes while unassisted by a walker or another person (the use of a cane is allowed).*
5. Mini Mental State Examination>= 21
6. At least three hours in-between regular medication intakes to allow for stable testing time.*
7. Self-reported FOG with a severity of at least 1 FOG episode per day, based on items 1 and 2 of the New Freezing of Gait Questionnaire, irrespective of FOG occurring ON- or OFF-medication.*
8. Stable medication scheme for at least 7 days before enrollment.

Exclusion Criteria:

1. Participation in another clinical intervention study*
2. Acute musculoskeletal or other neurological, psychiatric, or cardiovascular conditions affecting gait or any other medical condition which, in the opinion of the investigator, may prevent the participant from completing the protocol in full
3. Unable to adhere to assessment procedures leading to missing or unusable data, as determined by the investigators
4. Not a stable medication scheme for at least 7 days before the assessment.*
5. Occurrence of any of the following within 3 months prior to informed consent:

   * Orthopedic surgery of the lower extremity
   * Myocardial infarction
   * Hospitalization for unstable angina
   * Coronary artery bypass graft
   * Percutaneous coronary intervention
   * Implantation of a cardiac resynchronization therapy device
   * Implantation of deep brain stimulation
6. Substance abuse that may interfere with the patient's compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's Disease who self-report to experience FOG more than once a day.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Power spectral density (Watts/hertz) of beta frequencies | During walking protocol (duration 15-20 minutes)
  The averaged power spectral density (PSD) of the beta (12-25 Hz) frequency band measured over the motor cortices during freezing of gait (FOG) episodes compared to typical gait performance in the same individual with Parkinson's disease as measured during different walking trajectories in the home setting.

SECONDARY OUTCOMES:
Power spectral density (Watts/hertz) of theta frequencies bands | During walking protocol (duration 15-20 minutes)
  The averaged power spectral density (PSD) of the theta (4-7 Hz) frequency band measured over the prefrontal cortices during freezing of gait (FOG) episodes compared to typical gait performance in the same individual with Parkinson's disease as measured during different walking trajectories in the home setting.
Cross-frequency coupling between beta and theta frequency bands | During walking protocol (duration 15-20 minutes)
  The averaged cross-frequency coupling (CFC) between the beta (12-25 Hz) and theta (4-7 Hz) frequency bands as measured over the motor and prefrontal cortices during freezing of gait (FOG) episodes compared to typical gait performance in the same individual with Parkinson's disease as measured during different walking trajectories in the home setting.
Power spectral density (Watts/hertz) and cross-frequency coupling (CFC) of beta and theta frequencies bands over other cortical areas. | During walking protocol (duration 15-20 minutes)
  The averaged power spectral density (PSD) of the beta (12-25 Hz) and theta (4-7 Hz) frequency band measured over other cortical areas (prefrontal, motor, temporal, parietal, visual) during freezing of gait (FOG) episodes compared to typical gait performance in the same individual with Parkinson's disease as measured during different walking trajectories in the home setting.

OTHER OUTCOMES:
Power spectrum density and cross-frequency coupling in ON medication state | During walking protocol (duration 15-20 minutes)
  Comparing the PSD/CFC of the primary and secondary outcomes averaged across all FOG episodes to typical gait performance during optimal ON medication state (1 hour post-medication intake)
Power spectrum density and cross-frequency coupling in OFF medication state | During walking protocol (duration 15-20 minutes)
  Comparing the PSD/CFC of the primary and secondary outcomes averaged across all FOG episodes to typical gait performance during the practically defined OFF medication state (after minimal 12 hours overnight withdrawal).
Comparing the Power spectrum density and cross-frequency coupling in ON and OFF medication state | During walking protocol (duration 15-20 minutes)
  Comparing the PSD/CFC averaged across all FOG episodes compared to typical gait performance between OFF and ON medication states
Comparing the Power spectrum density and cross-frequency coupling between different FOG manifestations | During walking protocol (duration 15-20 minutes)
  Comparing the averaged PSD/CFC between the different FOG manifestations (Akinetic vs. Kinetic FOG trembling vs. Kinetic non-trembling vs. Kinetic-festination) in the ON and OFF medication states.

CONTACTS AND LOCATIONS:
Overall Officials: Moran Gilat, PhD, Principal Investigator — KU Leuven
Locations (1):
- Department of rehabilitation sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The datasets could be made available under restricted access after publication of the results, following ethical approval and a data-transfer agreement. GDPR and privacy regulations will be adhered to.